CLINICAL TRIAL: NCT00575861
Title: Evaluation of Additive Effects of Zileuton to Advair on Total Exhaled, Bronchial, and Alveolar Nitric Oxide in Asthmatics
Brief Title: Zileuton and Exhaled Nitric Oxide in Asthmatics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gelb, Arthur F., M.D. (Individual)
Responsible Party: Arthur F. Gelb MD, Arthur F. Gelb Medical Corporation
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2000; Critical Therapeutics, Inc.
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-12

CONDITIONS: Asthma
Keywords: asthma; nitric oxide gas exchange; lung function
MeSH Terms: conditions — Asthma | interventions — zileuton

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Advair 250/50 (baseline) fluticasone/salmeterol 250/50
  Interventions: Drug: zileuton

INTERVENTIONS:
Drug: zileuton — zileuton (Zyflo) 600mg qid for 2hr and for 30 days
  Other Names: zyflo

SUMMARY:
Evaluate the additive role of zileuton 600mg qid to clinically stable asthmatics on Advair 250/50 bid. Since asthma is an endogenous inflammatory disease there usually is increased total exhaled, bronchial and alveolar nitric oxide which are markers of eosinophilic driven pathways of inflammation. The addition of zileuton which is a leukotriene synthesis inhibitor by itself or together with inhaled corticosteroids should reduce nitric oxide gas exchange.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Moderate to severe persistent asthmatics
* Clinically stable X 6 weeks on Advair 250/50 bid for at least 12 months

Exclusion Criteria:

* No leukotriene synthesis inhibitors or receptor antagonists for 6 weeks

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
nitric oxide gas exchange including total exhaled nitric oxide, bronchial and alveolar nitric oxide | 2 hr to 1 month

SECONDARY OUTCOMES:
expiratory spirometry and asthma symptom Juniper score | 2 hr to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Arthur F Gelb Medical Corporation, Lakewood, California, United States

REFERENCES:
- [Background] Gelb AF, Flynn Taylor C, Shinar C, et al. Additive role of zileuton on total exhaled, bronchial, alveolar nitric oxide in non-atopic moderate to severe persistent asthmatics on fluticasone 250/salmeterol 50. Chest 2006;130:163S
- [Background] Gelb AF, Flynn Taylor C, Shinar CM, Gutierrez C, Zamel N. Role of spirometry and exhaled nitric oxide to predict exacerbations in treated asthmatics. Chest. 2006 Jun;129(6):1492-9. doi: 10.1378/chest.129.6.1492. PMID 16778266
- [Background] Gelb AF, Taylor CF, Nussbaum E, Gutierrez C, Schein A, Shinar CM, Schein MJ, Epstein JD, Zamel N. Alveolar and airway sites of nitric oxide inflammation in treated asthma. Am J Respir Crit Care Med. 2004 Oct 1;170(7):737-41. doi: 10.1164/rccm.200403-408OC. Epub 2004 Jun 30. PMID 15229098
- [Derived] Gelb AF, Taylor CF, Simmons M, Shinar C. Role of add-on zileuton on total exhaled, large airway, and small airway/alveolar nitric oxide in moderate-severe persistent adult asthmatics on fluticasone 250 microg/Salmeterol 50 microg. Pulm Pharmacol Ther. 2009 Dec;22(6):516-21. doi: 10.1016/j.pupt.2009.05.003. Epub 2009 May 23. PMID 19467341